CLINICAL TRIAL: NCT02479152
Title: The Haemodynamic Effects of Mechanical Standard and Active External Chest Compression-decompression During Out-of-hospital Cardiopulmonary Resuscitation
Brief Title: The Haemodynamic Effects of Mechanical Standard and Active Chest Compression-decompression During Out-of-hospital CPR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Physio-Control (Industry)
Collaborators: GE Healthcare (Industry)
Responsible Party: Principal Investigator, Lars Wik, MD, PhD, Ullevaal University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Protocol ID 11, March 2015
Record Dates: First submitted 2015-04-13; First posted 2015-06-24 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Cardiac Arrest
Keywords: Mechanical CPR; Hemodynamics
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LUCAS 2 AD (Active Comparator): LUCAS 2 AD will be used for CPR
  Interventions: Device: LUCAS2 AD
- LUCAS2 (Other): LUCAS2 will be used for CPR
  Interventions: Device: LUCAS2 AD

INTERVENTIONS:
Device: LUCAS2 AD — LUCAS™ 2AD with compressions like the standard LUCAS™ 2 but added decompressions above the initial start position.

SUMMARY:
The aim of this randomized out-of-hospital cardiopulmonary resuscitation study is to investigate haemodynamics generated by the standard mechanical external chest compression device (LUCAS™ 2) compared to a new version generating chest compressions and active decompression above the initial starting position of the suction cup (LUCAS™ 2AD).

DETAILED DESCRIPTION:
Based on randomization patients will receive standard or active compression decompression chest compression and the haemodynamic effects will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Unexpected adult out-of-hospital non-traumatic cardiac arrest where an attempt of resuscitation is considered appropriate in:
* Patients 18 years or older

Exclusion Criteria:

* Traumatic cardiac arrest
* Age believed to be less than 18 years
* Known pregnancy
* Victim not to be resuscitated (DNR orders)
* Internals in prison
* Included once in the study already
* To Small/Large patients
* Sustained ROSC occurring before the LUCAS™ 2 or LUCAS™ 2-AD can be applied to the patient, such that further CPR is not needed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Hemodynamics measured as EtCO2 | During 30 minutes of CPR

SECONDARY OUTCOMES:
Intra arterial blood pressures, | During 30 minutes of CPR
Oximetry, | During 30 minutes of CPR
ROSC (Return of spontaneous circulation) | During CPR
safety | During 30 minutes of CPR

CONTACTS AND LOCATIONS:
Overall Officials: Lars Wik, MD, PhD, Principal Investigator — Oslo Universitetssykehus. Ullevål, Norway.
Locations (1):
- Oslo University hospital, Oslo, Norway

REFERENCES:
- [Derived] Berve PO, Hardig BM, Skalhegg T, Kongsgaard H, Kramer-Johansen J, Wik L. Mechanical active compression-decompression versus standard mechanical cardiopulmonary resuscitation: A randomised haemodynamic out-of-hospital cardiac arrest study. Resuscitation. 2022 Jan;170:1-10. doi: 10.1016/j.resuscitation.2021.10.026. Epub 2021 Oct 25. PMID 34710550